CLINICAL TRIAL: NCT00741715
Title: A Multicenter, Randomized, Placebo-controlled, "Factorial" Design, 12-month Study to Evaluate the Efficacy and Safety of AVE5530 25 mg/Day and 50 mg/Day Co-administered With All Registered Atorvastatin Strengths Ranging From 10 mg to 80 mg in Patients With Primary Hypercholesterolemia
Brief Title: Evaluation of Efficacy and Safety of AVE5530 Co-administered With Atorvastatin in Primary Hypercholesterolemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: AVE5530 in hypercholesterolemia was stopped due to insufficient efficacy
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC6911
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Hypercholesterolemia
Keywords: primary hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (15):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental): AVE5530 25mg
  Interventions: Drug: AVE5530
- 3 (Experimental): AVE5530 50mg
  Interventions: Drug: AVE5530
- 4 (Active Comparator): atorvastatin 10mg
  Interventions: Drug: atorvastatin
- 5 (Experimental): atorvastatin 10mg + AVE5530 25mg
  Interventions: Drug: AVE5530; Drug: atorvastatin
- 6 (Experimental): atorvastatin 10mg + AVE5530 50mg
  Interventions: Drug: AVE5530; Drug: atorvastatin
- 7 (Active Comparator): atorvastatin 20mg
  Interventions: Drug: atorvastatin
- 8 (Experimental): atorvastatin 20mg + AVE5530 25mg
  Interventions: Drug: AVE5530; Drug: atorvastatin
- 9 (Experimental): atorvastatin 20mg + AVE5530 50mg
  Interventions: Drug: AVE5530; Drug: atorvastatin
- 10 (Active Comparator): atorvastatin 40mg
  Interventions: Drug: atorvastatin
- 11 (Experimental): atorvastatin 40mg + AVE5530 25mg
  Interventions: Drug: AVE5530; Drug: atorvastatin
- 12 (Experimental): atorvastatin 40mg + AVE5530 50mg
  Interventions: Drug: AVE5530; Drug: atorvastatin
- 13 (Active Comparator): atorvastatin 80mg
  Interventions: Drug: atorvastatin
- 14 (Experimental): atorvastatin 80mg + AVE5530 25mg
  Interventions: Drug: AVE5530; Drug: atorvastatin
- 15 (Experimental): atorvastatin 80mg + AVE5530 50mg
  Interventions: Drug: AVE5530; Drug: atorvastatin

INTERVENTIONS:
Drug: AVE5530 — oral administration once daily in the evening with dinner
  Arms: 11; 12; 14; 15; 2; 3; 5; 6; 8; 9
Drug: atorvastatin — oral administration once daily in the evening with dinner
  Arms: 10; 11; 12; 13; 14; 15; 4; 5; 6; 7; 8; 9
Drug: placebo — oral administration once daily in the evening with dinner
  Arms: 1

SUMMARY:
The present study is assessing the efficacy and safety of AVE5530 (25mg and 50mg) co-administered with all approved doses of atorvastatin in a double-blind comparison with placebo, AVE5530 alone and atorvastatin alone in the management of patients with primary hypercholesterolemia. The main objective is to evaluate the effects of the association AVE5530+atorvastatin on LDL-C level reduction after 12 weeks of treatment. The effects of AVE5530+atorvastatin on other lipid parameters will be assessed as secondary objectives

DETAILED DESCRIPTION:
The study will include a 2 week pre-randomization placebo lead-in phase. There will be a 12- week double-blind treatment period for both components AVE5530 and atorvastatin, followed by a 40-week period with maintenance of double-blind design for AVE5530 component and open label for atorvastatin component transitioning at 20 mg for all patients with subsequent titration, if necessary, based on regular LDL-cholesterol monitoring. The treatment period can be variably extended up to approximately 18 months with double-blind for AVE5530 component and open-label for atorvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Adults with high cholesterol levels either not receiving or willing and able to discontinue ongoing lipid-lowering therapy

Exclusion Criteria:

* LDL-C levels > 250 mg/dL (6.48 mmol/L)
* Triglycerides levels > 350mg/dL (3.95 mmol/L)
* Conditions / situations such as:

  * presence of any clinically significant uncontrolled endocrine disease known to influence lipids levels
  * Active liver disease
  * High estimated risk of Coronary Heart Disease
  * Recent history of congestive heart failure , of unstable angina pectoris, myocardial infarction, coronary bypass surgery or angioplasty, or Unstable or severe peripheral artery disease
  * Positive test for Hepatitis B surface antigen and/or Hepatitis C antibody or Known to be Human Immunodeficient Virus (HIV) positive
* Pregnant or breast-feeding women,
* Women of childbearing potential not protected by effective contraceptive method of birth control (including oral contraceptives) and/or who are unwilling or unable to be tested for pregnancy prior to exposure to the Investigational Product
* Hypersensitivity to any component of atorvastatin
* Concurrent administration of Cytochrome P450 3A4 inhibitors (e.g. cyclosporine, erythromycin, clarithromycin, and azole antifungals) should be avoided as increasing the risk of myopathy with atorvastatin

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1736 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in calculated LDL-C | At week 12

SECONDARY OUTCOMES:
Percent change from baseline in calculated LDL-C | At 6 months and 12 months
Percent change from baseline in total cholesterol, HDL-C, TG, Apo-A1, Apo-B and CRP | At week 12, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Davidson Michael, MD, Principal Investigator — Radiant Research - 515 North State Street Suite 2700 Chicago Illinois (US)
Locations (2):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, San Juan, Puerto Rico